CLINICAL TRIAL: NCT05483309
Title: Feasibility Study of the Clinical and Cost-effectiveness of Contemporary Diagnostics for Patients With Suspected Hospital-Acquired Pneumonia (HAP).
Brief Title: Feasibility Study of Contemporary Diagnostics for Patients With Suspected Hospital-Acquired Pneumonia.
Acronym: HAP-FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UoL001676
Record Dates: First submitted 2022-07-05; First posted 2022-08-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-01

CONDITIONS: Hospital-acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Diagnostic Treatment Regimen 1 (Experimental): Patients will receive a chest x-ray and their sputum sample will be analysed using the FilmArray Pneumonia Panel.
  Interventions: Diagnostic Test: FilmArray Pneumonia Panel
- Diagnostic Treatment Regimen 2 (No Intervention): Patients will receive a chest x-ray and their sputum sample will not be analysed using the FilmArray Pneumonia Panel.
- Diagnostic Treatment Regimen 3 (Experimental): Patients will receive a CT scan and their sputum sample will be analysed using the FilmArray Pneumonia Panel.
  Interventions: Diagnostic Test: CT scan; Diagnostic Test: FilmArray Pneumonia Panel
- Diagnostic Treatment Regimen 4 (Experimental): Patients will receive a CT scan and their sputum sample will not be analysed using the FilmArray Pneumonia Panel.
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Patients receive a CT scan
  Arms: Diagnostic Treatment Regimen 3; Diagnostic Treatment Regimen 4
Diagnostic Test: FilmArray Pneumonia Panel — The FilmArray Pneumonia Panel is used to analysis the patient's sputum sample for the cause of the hospital acquired pneumonia
  Arms: Diagnostic Treatment Regimen 1; Diagnostic Treatment Regimen 3

SUMMARY:
Hospital-Acquired Pneumonia (HAP) is a severe lung infection that develops while a patient is in hospital. We aim to design a trial to see if modern diagnostic investigations can safely improve outcomes for patients suspected of HAP.

Currently, doctors use chest x-rays to make the diagnosis, but these are difficult to interpret and a third of patients suspected of HAP receive antibiotics inappropriately. Patients are concerned about misdiagnosis and a solution might be to replace the chest x-ray with a CT scan since these show the lungs in more detail.

Once a diagnosis of HAP is made, doctors would like to identify the bacteria or viruses responsible. However, current tests are too slow to determine the initial treatment, so guidelines suggest we cover a range of possibilities with two extended spectrum antibiotics. Patients tell us they are concerned, because these antibiotics increase the risk of severe side effects and promote antibiotic resistance. The BIOFIRE® FILMARRAY® pneumonia panel (FAPP) is a new test that can identify the cause of HAP quickly. If we can determine the best way to use the FAPP, we can give antibiotics more effectively and slow the development of antimicrobial resistance.

We will conduct a feasibility study to inform the design of a fully powered trial to discover whether using CT scans or the FAPP, or both together, helps improve antibiotic use and patient recovery whilst being cost effective.

We will interview some participants and staff about how the trial is working so that we can improve the design. We will list the costs associated with HAP so we can design a cost effectiveness evaluation for the definitive trial. We will use patient samples to investigate immune and inflammation related processes to better understand why some people develop HAP and why some become particularly unwell.

ELIGIBILITY:
Inclusion Criteria:

Stage 1:

* Age ≥ 18 years
* Suspected HAP*

For the purposes of this study, HAP is defined as per the BTS and FDA definitions i.e. pneumonia which develops 48 hours after an admission to hospital for an alternative diagnosis; or a new presentation to hospital with pneumonia in a patient who has been discharged from an overnight stay in hospital within the last 10 days.

Stage 2:

* The clinician intends to treat the patient for HAP or a hospital acquired respiratory tract infection (RTI).
* A sputum sample has been obtained before 2nd dose of antibiotic.

Exclusion Criteria:

Stage 1:

* Already received a chest X-ray to confirm suspected HAP diagnosis
* Diagnosis or suspected diagnosis of ventilator acquired pneumonia
* Intention to palliate rather than cure
* Interventions cannot be completed before administration of second antibiotic dose*
* Cannot be randomised to low-dose, non-contrast CT scan on clinical grounds e.g. strong suspicion of PE**
* Pregnancy***
* Previous study participation (patients with second of third episodes of HAP will not be re-recruited)

In the circumstance where a patient is diagnosed with HAP whist receiving antibiotics for a non-respiratory infection e.g. cellulitis or UTI, if the HAP diagnosis leads to a change in the antibiotic prescription to cover the HAP then that patient will be eligible for recruitment. However, if the diagnosis of HAP does not result in a change in antibiotic then the patient is not eligible.

A non-contrast, low-dose thoracic CT scan is an inappropriate test for a PE and if that is high in the differential diagnosis then tick yes here.

A urine pregnancy test is required as part of routine care prior to a chest X-ray or CT scan. If the test reveals the patient is pregnant, they will not be eligible for the study as they will be unable to receive a CT scan as part of this study. Pregnancy tests are not required at future time points.

Stage 2:

- Following the CXR or CT the clinician decides not to treat with antibiotics for either HAP or a hospital acquired RTI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of a full-scale Randomised Controlled Trial (RCT) comparing different diagnostic dynamic treatment regimens (DTRs) in adult patients suspected of HAP. | Screening and randomisation (1 year); follow up (3 months); end of study analysis (9 months).
  Rate of recruitment; proportion screened that meet eligibility criteria; proportion eligible that consent and where they present; proportion consented and randomised that complete study pathway as per protocol; proportion consented and randomised that withdraw from trial intervention or follow up.

SECONDARY OUTCOMES:
Estimate population statistics for each DTR - Time to clinical cure | Day 90
  Time to clinical cure, defined as the number of days from baseline when there is a combination of resolution of signs and symptoms present at enrolment and improvement or lack of progression of radiological signs.
Estimate population statistics for each DTR - Antibiotic usage | Day 90
  Antibiotic usage for the HAP episode
Estimate population statistics for each DTR - Change to Quality of Life | Baseline, day 10, 28 and 90
  Change of quality of life using the EQ-5D-5L measure
Estimate population statistics for each DTR - Length of hospital stay | Day 90
  Length of hospital stay post HAP diagnosis.
Estimate population statistics for each DTR - Mortality | Day 14, 28 and 90
  We will evaluate the best way to record this by analysing: in-hospital mortality, survival at three timepoints.
Estimate number of eligible patients and the pattern of their presentation. | At end of study (15 months)
  Hospital/ward type, time of day/day of week.
Estimate rates of successful follow up. | At end of study (15 months)
  Participants who attend 28 day visit and complete the post discharge indirect cost survey at 90 days.
Estimate rates of completion of questionnaires. | At end of study (15 months)
  EQ5D5L, CAP-sym, economic evaluation.
Test the web-based randomisation process and incorporate clinical and researcher feedback. | During qualitative analysis throughout the study (up to 15 months)
  Qualitative conclusions based on staff focus groups.
Perform a costing analysis of HAP to inform the cost-effectiveness analysis for any definitive trial. | At end of study (15 months)
  Summary statistics for numbers and types of costs with comparison between DTRs.
Assess human factors involved in delivery of the study and how the different diagnostic tests influence clinical decision making by conducting qualitative interviews and focus groups with healthcare workers and researchers. | During qualitative analysis throughout the study (up to 15 months)
  Qualitative conclusions based on staff focus groups.
Evaluate willingness of clinicians to recruit to the study. | During qualitative analysis throughout the study (up to 15 months)
  Qualitative conclusions based on staff focus groups.
Evaluate willingness of potential participants or their consultees to be recruited. | During qualitative analysis throughout the study (up to 15 months)
  Qualitative conclusions based on participant and carer interviews.
Evaluate adherence to antibiotic guidelines and study protocol. | At end of study (15 months)
  Summary statistics relating to antibiotic use in the pilot study with a comparison between the DTRs.
Assess the study participant and carer experience of participating in the study. | During qualitative analysis throughout the study (up to 15 months)
  Qualitative interviews.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Manchester University NHS Foundation Trust, Manchester
  - Lancashire teaching hospitals NHS Foundation Trust, Preston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shafiqa N, Aston S, Howard A, Turtle L, Abrams S, Young B, Sherratt F, Alvarez Nishio A, Wilshaw S, Jones AP, Wootton DG. HAP-FAST: a feasibility study incorporating qualitative, mechanistic and costing sub-studies alongside a randomised pilot trial comparing chest x-ray to low-dose CT scan and empirical antibiotics to antibiotics guided by the BIOFIRE(R) FILM ARRAY(R) pneumonia plus panel in adults with suspected non-ventilator-associated hospital-cquired pneumonia. BMJ Open. 2024 Jul 4;14(7):e088490. doi: 10.1136/bmjopen-2024-088490. PMID 38964799